CLINICAL TRIAL: NCT06144255
Title: Phase 1, Dose-Dependent Effect of Intranasal Insulin in Humans Using Functional MRI
Brief Title: Dose-Dependent Effect of Intranasal Insulin in Humans Using Functional Magnetic Resonance Imaging (fMRI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Florian Schmitzberger (Other)
Responsible Party: Sponsor-Investigator, Florian Schmitzberger, Instructor in Emergency Medicine, University of Michigan
Organization: University of Michigan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00230748
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Healthy
Keywords: Healthy Participants; Intranasal Insulin; Functional Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Each volunteer will have 3 study visits, receiving a different study dose at each visit in randomized order as spelled out in the protocol.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intranasal insulin and placebo (Experimental): A total of 3 possible doses will be tested of insulin 0 units (u) (placebo (diluent), 500u, and 1000u. The order that participants will receive these doses will be in a random order.
  Interventions: Drug: Intranasal insulin

INTERVENTIONS:
Drug: Intranasal insulin — Enrolled Participants for this trial will come for 3 study visits. The doses will be administered in varying order: participants will be randomized to one six possible permutations of the intranasal study doses (0, 500, 1000 U) of intranasal insulin at each visit.
  Participants will undergo a fMRI scan before and after receiving intranasal doses. Additionally, participants will have blood samples taken.
  Other Names: HUMULIN R U-500

SUMMARY:
The purpose of this trial is to study the brain response using functional MRI (fMRI) before and after varying doses of insulin given through the nose. The magnetic resonance imaging uses a very strong magnet to produce images of participant's brain. It becomes a functional MRI when the study team looks at the activity within the brain (blood flow / change in metabolism).

DETAILED DESCRIPTION:
If cardiac arrest is not treated immediately, it causes sudden death. Intranasal insulin may be a way to prevent the brain injury that occurs after a cardiac arrest or other brain injury. Even when immediate treatment gets the heart beating again, many victims remain comatose and die later from brain injury. Nasal insulin reduces brain injury in animal experiments and has been used to try to improve brain degeneration in patients with Alzheimer's disease in doses up to 160 units.

ELIGIBILITY:
Inclusion Criteria:

* Participants in good health based on medical history, physical exam, and routine laboratory testing
* Female participants must have a negative urine pregnancy test or be surgically sterilized or postmenopausal. Criteria for menopause are surgical menopause (hysterectomy, oophorectomy) or age > 45 years with the absence of menses for greater than 12 months.
* Body mass index (BMI) between 18 kg/m2 and 35 kg/m2
* Willing and able to stay at the clinical research facility as required by the protocol
* Willing and able to comply with the investigational nature of the study and able to communicate well with investigators
* Ability to comprehend and willing to provide written informed consent in accordance with institutional and regulatory guidelines
* Ability to lie flat for a minimum of 2-hours

Exclusion Criteria:

* Known allergy to insulin.
* Preexisting diabetes.
* Current or previous use of diabetes medication or insulin.
* Any nasal disease or congestion that may interfere with intranasal drug absorption.
* Baseline hypoglycemia (blood glucose ≤ 65 milligrams per deciliter (mg/dL)) or hyperglycemia (blood glucose > 200 mg/dL) as evident from the screening labs.
* Active serious disease, such as liver disease, kidney disease, uncontrolled hypertension, clinically significant hypokalemia, and significant or unstable medical illness
* Treated with an investigational drug within 30 days.
* Individuals with inadequate venous access.
* Claustrophobic, uncontrollable shaking, or unable to lie still for a lengthy period.
* Any metals or implanted devices within the body.
* Any foreign metallic objects in the body.
* Females that are pregnant, trying to become pregnant, or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Change in Signal response using fMRI after administration of intranasal insulin | Baseline fMRI (approximately 30 minutes), fMRI Approximately 30 minutes (after insulin dose administration)
  Values of regions of interest in the fMRI will be calculated for all measures, including cerebral blood flow (CBF), at different used dosages and compared directly as well as with baseline-corrected CBF maps. The study team will determine if a significant difference at different dosages exists.

SECONDARY OUTCOMES:
Change in Blood Glucose (serum or point of care capillary) | Baseline (Immediately before drug administration), up to approximately 90 minutes (after drug dose)

CONTACTS AND LOCATIONS:
Overall Officials: Florian Schmitzberger, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No